CLINICAL TRIAL: NCT03576638
Title: An Open Label Phase 2 Study to Assess the Pharmacokinetics of the Accordion Pill Carbidopa-Levodopa Compared to Immediate Release Carbidopa-Levodopa in Patients With Parkinson's Disease
Brief Title: Study to Assess Pharmacokinetics of Accordion Pill Carbidopa-Levodopa Compared to Immediate Release Carbidopa-Levodopa in Parkinson's Disease Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Intec Pharma Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IN 18001; 2018-001209-95 (EudraCT Number)
Record Dates: First submitted 2018-06-25; First posted 2018-07-03 (Actual); Last update posted 2018-07-05 (Actual); Status verified 2018-06

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Carbidopa; Levodopa; carbidopa, levodopa drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sinemet (Active Comparator): Controlled Release 25/100
  Interventions: Drug: Sinemet CR 25Mg-100Mg Extended-Release Tablet
- AP CD/LD (Experimental)
  Interventions: Drug: Accordion Pill Carbidopa/Levodopa

INTERVENTIONS:
Drug: Accordion Pill Carbidopa/Levodopa — AP 50/500 TID days 2-7
  Other Names: AP-CD/LD
  Arms: AP CD/LD
Drug: Sinemet CR 25Mg-100Mg Extended-Release Tablet — 25/100 1.5 pills five times/day
  Other Names: Sinemet CR
  Arms: Sinemet

SUMMARY:
The purpose of this study is to assess the PK of AP-CD/LD given at dose of 50/500mg three times daily compared to CD/LD immediate release (Sinemet) 1.5 tablets of dose of 25/100 given 5 times per day in Parkinson's Disease patients.

DETAILED DESCRIPTION:
An open label, non randomized crossover phase 2 study to assess the PK of AP-CD/LD given at dose of 50/500mg three times daily compared to CD/LD immediate release (Sinemet) 1.5 tablets of dose of 25/100 given 5 times per day in Parkinson's Disease patients. The study will have a screening period followed by an overnight stay in clinic where Immediate release CD/LD (Sinemet) will be administered five times, approximately every three hours. At specified intervals, blood will be drawn for PK testing. On Days 2-7, subjects will be treated at home with AP CD/LD three times/day, approximately every five hours. Day 8 will be overnight stay in clinic for PK study. AP CD/LD 500mg TID will be dispensed to subjects with specified timelines for PK assessment. Each subject will return to clinic on day 15 for a safety followup visit.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of PD consistent with UK Brain Bank Criteria
2. Stable dose of levodopa/carbidopa IR for at least 4 weeks prior to entry; taking at least 4 doses of IR levodopa during waking hours, and total daily dose of at least 400mg prior to initial screening
3. Stable on all anti-PD medications for 30 days prior to screening. COMT inhibitors are held prior to PK studies on day 1 through day 8

Exclusion Criteria:

1. Atypical or secondary parkinsonism
2. clinically significant cardiac, pulmonary, hepatic, or renal disease or other condition which contraindicates participation in judgement of investigator
3. severe dyskinesia as assessed by PI
4. significant cognitive impairment
5. Clinically significant psychiatric illness in opinion of PI
6. history of small bowel or gastric surgery (including PEG-J placement for Duopa/Duodopa) or bowel obstruction, diagnosis of small bowel narrowing, diagnosis of Crohn's disease, frequent nausea or emesis regardless of etiology, and symptomatic gastroparesis.
7. History of GI pathology of clinical significance as determined by PI
8. Allergy to study drug or Yellow Dye #5 (tartrazine)
9. Unable to swallow large pills
10. Active GERD and regular use of PPIs
11. Women who are pregnant or nursing or are of childbearing potential who are not willing to use a medically acceptable method of contraception

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2018-07 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Variability in plasma levodopa concentration | Pk blood sampling to be performed time 0 and every 30 minutes for 16 hours and again at 24 hours on days 1 and 8.
  as assessed by levodopa fluctuation index (comparison of AP-CD/LD to IR-CD/LD

SECONDARY OUTCOMES:
Variability in plasma levodopa concentration | Pk blood sampling to be performed time 0 and every 30 minutes for 16 hours and again at 24 hours on days 1 and 8.
  as assessed by Coefficient of variation (CV) (comparison of AP-CD/LD to IR-CD/LD)